CLINICAL TRIAL: NCT07279467
Title: Study of Oral Food Challenge Biomarkers (CoFAR-15)
Brief Title: Study of Oral Food Challenge Biomarkers (SAFER)
Acronym: SAFER
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Consortia for Food Allergy Research (CoFAR) (Unknown); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT CoFAR-15
Record Dates: First submitted 2025-09-30; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Allergy
Keywords: Food Allergy; Peanut Allergy; Oral Food Challenge; CoFAR-15; SAFER; Biomarkers
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Food Challenge Cohort: Approximately 500 children and adolescent participants between the ages of 1-17 years who are suspected of having an allergy to peanut will be asked to complete a Peanut Oral Food Challenge. An individual's participation in this study will consist of screening for eligibility and an oral food challenge visit, which may occur on the same day or up to 28 days apart.
  Interventions: Drug: Oral Food Challenge (OFC): Peanut Protein

INTERVENTIONS:
Drug: Oral Food Challenge (OFC): Peanut Protein — Peanut protein flour will be used in the OFC procedure. The maximum cumulative dose of peanut protein for completion of the oral food challenge (OFC) is 6043 mg. Participants aged 3 years or younger are not required to receive the final 2000 mg dose to complete the OFC; however, it may be administered at the discretion of the investigator if considered clinically relevant and safe.
  Other Names: OFC

SUMMARY:
This is a multi-center, mechanistic study. It is designed to learn more about signs in the body, called biomarkers, that might show if someone will have a reaction to peanut during a feeding test. The trial will enroll children ages 12 months to17 years old who are suspected of having an allergy to peanut.

The primary objective is to identify a biomarker (or a combination of biomarkers) that will predict oral food challenge (OFC) (feeding test) results for participants with suspected peanut allergy.

DETAILED DESCRIPTION:
The SAFER study is a multi-center, mechanistic study designed to identify biomarkers that can predict the outcome of a participant's reactions to a peanut oral food challenge. Participants aged 12 months to 17 years with suspected peanut allergy will complete an oral food challenge to peanut. The accrual goal of the study is to reach a minimum of 500 participants who complete the oral food challenge and provide blood needed to assess biomarkers. Recruitment may continue beyond 500 to ensure there are at least 350 reactors (i.e., participants who experience dose-limiting symptoms during the OFC) and 100 non-reactors. Recruitment will aim to achieve approximate balance across three age groups: 12-47 months, 4-11 years, and 12-17 years.

An initial screening visit will be conducted to evaluate eligibility and collect the biomarkers prior to the oral food challenge. The food challenge can take place on the same day as screening or within 4 weeks of the screening visit.

During participation, clinical assessments will be conducted, questionnaires completed, and biological samples collected from the participant before, during, and after the challenge.

After the food challenge and the safety monitoring period is completed, the participant will have completed participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or guardian must be able to understand and provide written informed consent and participant must be able to understand and provide assent (if applicable)
2. Are 12 months - 17 years of age during Screening.
3. Are sensitized to peanut, as demonstrated by one of the following:

   a. A participant-reported reaction to peanut (at any time) deemed by the investigator to be consistent with an IgE-mediated reaction and one of the following within the past 12 months

   i. Positive Skin Prick Test (SPT) to peanut (wheal diameter that is ≥ 3mm larger than saline control) ii. Positive peanut-specific IgE (sIgE; ≥ 0.10 kUA/L) determined by ImmunoCap

   b. An Ara h 2 sIgE ≥ 1.0 kUA/L, measured within the past 12 months
4. Are currently avoiding peanut

Exclusion Criteria:

1. Are pregnant
2. Are currently receiving treatment or have received treatment within the prior 2 years for peanut allergy
3. Have a history of life-threatening anaphylaxis to peanut, defined as neurological compromise or requiring intubation
4. Have received treatment with dupilumab/Dupixent® within the prior 2 years, OR treatment with omalizumab/Xolair®, other biologics, or systemic immunomodulatory agents within the prior year
5. Inability to comply with the required aspects of the study protocol
6. Have past or current medical conditions or findings from the physical examination, not already listed, that, in the judgment of the site investigator, may pose additional risks related to participation in the study, interfere with the participant's ability to comply with study requirements, or impact the quality or interpretation of the study data
7. Have been treated with oral steroid or beta blockers within 14 days of the Oral Food Challenge (OFC)
8. Are unable to discontinue medications, as specified in the Protocol CoFAR-15 MOP, for the minimum wash-out periods prior to Skin Prick Test (SPT) or OFC
9. Have poorly controlled atopic dermatitis (AD) at Screening, per the PI's discretion
10. Have poorly controlled or severe asthma/wheezing at Screening, as defined as experiencing or including any of the following:

    1. Meeting the Global Initiative for Asthma (GINA) criteria for uncontrolled asthma
    2. History of two or more systemic corticosteroid courses within six months of Screening or one course of systemic corticosteroids within three months of Screening to treat asthma/wheezing;
    3. Prior intubation/mechanical ventilation for asthma/wheezing;
    4. One hospitalization or ED visit for asthma/wheezing within six months of Screening;
    5. Forced expiratory volume in one second (FEV1) <80% of predicted or FEV1/forced vital capacity (FVC) <75% of predicted, with or without controller medications (only for participants who are aged seven years or older and are able to perform spirometry);
    6. Inhaled corticosteroid (ICS) dosing of >500 mcg daily fluticasone (or equivalent ICS based on the CoFAR Inhaled Corticosteroid Equivalency Tables MOP)
11. Refuse blood sample collection during Screening
12. The SPT performed during Screening is negative to peanut allergen without dilution (wheal diameter that is < 3mm larger than saline control).

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 500 participants with suspected peanut allergy, 12 months to 17 years of age
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative Reactive Dose (CRD) Threshold | OFC Visit on Day 1
  The cumulative quantity of peanut protein consumed during an oral food challenge at which dose-limiting symptoms occur, categorized as: 3-143 mg (low threshold); 443-1043 mg (medium threshold); 2043-highest cumulative, age-dependent dose (high threshold); or no reaction.
  The maximum cumulative dose of peanut protein for completion of the oral food challenge (OFC) is 4043 mg for participants aged 1 to 3 years and 6043 mg for participants aged 4 to 17 years. Participants ≤3 years are not required to receive the final 2000mg dose to complete the OFC, however, it may be administered at the discretion of the investigator if considered clinically relevant and safe.
Binary Reaction Status (reactor/non-reactor) to the oral food challenge (OFC) | OFC Visit on Day 1
  A Reactor is any participant who experiences dose-limiting symptoms at or prior to the highest cumulative, age-dependent OFC dose. A Non-reactor is any participant who does not experience dose-limiting symptoms during an OFC that is completed to the age-specific highest dose.

SECONDARY OUTCOMES:
All reported treatments during the oral food challenge (OFC) or observational period. | OFC Visit on Day 1
  Any treatments used to resolve dose-limiting symptoms in response to the OFC, including during and after the OFC, will be summarized descriptively for participants who had at least 1 dose of peanut protein during the OFC (including those that started but did not fully complete the OFC).
All adverse events experienced during the OFC or observation period. | OFC Visit on Day 1
  Any adverse events, defined as severe dose-limiting symptoms that are related to the OFC, that are experienced during and after the OFC will be summarized descriptively in participants who had at least 1 dose of peanut protein during the OFC (including those that started but did not fully complete the OFC).
All symptoms reported during the OFC or observation period. | OFC Visit on Day 1
  All OFC symptoms (i.e. including those that do not meet definition of an adverse event) experienced during the OFC or after the OFC will be summarized descriptively in participants who had at least 1 dose of peanut protein during the OFC (including those that started but did not fully complete the OFC).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, M.D., Study Chair — Johns Hopkins Children's Center: Department of Allergy & Immunology; Supinda Bunyavanich, M.D., M.P.H., M.Phil., Study Chair — Icahn School of Medicine at Mount Sinai: Department of Pediatrics Allergy & Immunology; Charles Schuler, M.D., Study Chair — The University of Michigan: Division of Allergy and Clinical Immunology
Locations (10):
- United States (10):
  - Arkansas Children's Hospital Research Institute: Department of Pediatrics, Allergy & Immunology, Little Rock, Arkansas
  - Stanford School of Medicine: Sean N. Parker Center for Allergy & Asthma Research, Palo Alto, California
  - Northwestern University Feinberg School of Medicine: Allergy Division, Chicago, Illinois
  - Johns Hopkins Children's Center: Department of Allergy & Immunology, Baltimore, Maryland
  - Boston Children's Hospital: Allergy and Asthma Program, Boston, Massachusetts
  - The University of Michigan: Division of Allergy and Clinical Immunology, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai: Department of Pediatrics Allergy & Immunology, New York, New York
  - North Carolina Children's Hospital: Department of Pediatrics, Division of Allergy, Immunology and Rheumatology, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center: Division of Allergy and Immunology, Cincinnati, Ohio
  - Vanderbilt University Medical Center: Division of Pediatric Allergy, Immunology, and Pulmonary Medicine, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT/NIAID-funded awards and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/